CLINICAL TRIAL: NCT05300737
Title: Symptomatic Carotid Outcomes Registry With Multi-center Evaluation
Brief Title: Symptomatic Carotid Outcomes Registry
Acronym: SCORE
Status: Active, not recruiting | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Seemant Chaturvedi, Professor of Neurology, University of Maryland, Baltimore
Other Study IDs: 00088344-2
Record Dates: First submitted 2022-03-09; First posted 2022-03-29 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Carotid Stenosis; Ischemic Stroke; Transient Ischemic Attack
MeSH Terms: conditions — Carotid Stenosis; Ischemic Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Symptomatic carotid stenosis with low risk features: 50-99% symptomatic carotid stenosis with low clinical or radiologic risk features (see inclusion criteria) Patients will receive intensive medical therapy, including dual antiplatelet therapy, high potency statins, BP control, and lifestyle modification
  Interventions: Other: intensive medical therapy

INTERVENTIONS:
Other: intensive medical therapy — Dual antiplatelet therapy, high potency statins, HTN control, lifestyle modification

SUMMARY:
The purpose of this study is to build upon trials done over 30 years ago, which did not include statins, new antiplatelet agents, and newer antihypertensive medications. Since the landmark trials (NASCET, ECST), there have been new developments in medical stroke prevention, which creates a gap in knowledge. The aim of this study is to evaluate that clinical care with Intensive Medical Therapy (IMT) alone, the one year stroke rate in patients with symptomatic carotid stenosis and low risk clinical features will be <5%.

DETAILED DESCRIPTION:
This study will only be evaluating clinical care and no interventions will be done specifically for this research.

* Informed consent from patient or legally authorized representative.
* Participant survey/questionnaire completion at baseline, 6 and 12 months after enrollment
* All data collected will be entered into a secure research data registry created for this study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥40 years plus stroke or TIA ipsilateral to 50-99% ICA stenosis

In addition, patients must have at least one clinical or radiologic marker of reduced stroke risk

Clinical Reduced Stroke RISK:

1. Retinal ischemia only (amaurosis fugax, branch retinal artery occlusion (BRAO), central retinal artery occlusion (CRAO)
2. Female sex
3. Most recent stroke or TIA >1 week ago

Radiologic Reduced Stroke RISK:

1. Transcranial Doppler (TCD) study demonstrating lack of microembolic signals
2. Cross-sectional MRI plaque imaging demonstrating absence of intraplaque hemorrhage
3. For patients with TIA: brain MRI shows no DWI lesion

Exclusion Criteria:

Atrial fibrillation or other high-risk sources of cardiac embolism unless it is device detected AF only or duration <6 minutes

Alcohol and substance abuse within the prior 24 months

Clinically significant bleeding diathesis (platelet count <100K, prothrombin time >14 seconds)

Clear indication for therapeutic anticoagulation (for example, DVT or pulmonary embolism within past 3 months)

Left ventricular ejection fraction <20%

Known allergy or intolerance to aspirin or clopidogrel

Life expectancy less than 12 months

Moderate/severe dementia (Mini-mental or MOCA score <22

Modified Rankin score of >4

Nonatherosclerotic cause of carotid stenosis

Most recent symptomatic event >180 days from the time of enrollment

-

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with 50-99% symptomatic carotid stenosis and low risk clinical or radiologic features
Sampling Method: Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Ischemic stroke | within 12 months
  ipsilateral to carotid stenosis, with radiologic confirmation

SECONDARY OUTCOMES:
Myocardial infarction | within 12 months
  ECG will be performed for suspected myocardial infarction and will be diagnosed if appropriate ST changes and confirmation with troponin measurements

CONTACTS AND LOCATIONS:
Overall Officials: Seemant Chaturvedi, MD, Principal Investigator — School of Medicine, University of Maryland
Locations (18):
- United States (11):
  - Hartford Hospital, Hartford, Connecticut
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - University of Rochester, Rochester, New York
  - Rhode Island Hospital, Providence, Rhode Island
  - Baylor Medicine, Houston, Texas
- Canada (7):
  - Calgary Health Sciences Center, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, MN
  - Northern Ontario School of Medicine, Greater Sudbury, Ontario
  - Western University/London Health Sciences Center, London, Ontario
  - CHUM, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] King A, Markus HS. Doppler embolic signals in cerebrovascular disease and prediction of stroke risk: a systematic review and meta-analysis. Stroke. 2009 Dec;40(12):3711-7. doi: 10.1161/STROKEAHA.109.563056. Epub 2009 Oct 22. PMID 19850894
- [Result] Chaturvedi S. Treatment of a hot carotid: More fuel is needed to clarify the best treatments. Neurol Clin Pract. 2018 Dec;8(6):466-467. doi: 10.1212/CPJ.0000000000000561. No abstract available. PMID 30588374
- [Result] Saba L, Saam T, Jager HR, Yuan C, Hatsukami TS, Saloner D, Wasserman BA, Bonati LH, Wintermark M. Imaging biomarkers of vulnerable carotid plaques for stroke risk prediction and their potential clinical implications. Lancet Neurol. 2019 Jun;18(6):559-572. doi: 10.1016/S1474-4422(19)30035-3. Epub 2019 Apr 4. PMID 30954372
- [Result] Rothwell PM, Eliasziw M, Gutnikov SA, Warlow CP, Barnett HJ; Carotid Endarterectomy Trialists Collaboration. Endarterectomy for symptomatic carotid stenosis in relation to clinical subgroups and timing of surgery. Lancet. 2004 Mar 20;363(9413):915-24. doi: 10.1016/S0140-6736(04)15785-1. PMID 15043958